CLINICAL TRIAL: NCT05029778
Title: Efficacy L-arginine + L-citrulline as a Dietary Supplement vs Placebo for Weight Gain in Fetus With a Decrease in Their Growth Curve in the Third Trimester of Pregnancy
Brief Title: Arginine + Citrulline as a Supplement for Weight Gain in Fetus With a Decrease in Their Growth Curve
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jorge Bravo Rubio, Fetal and maternal medicine, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 097/20
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Fetal Growth Retardation
Keywords: L-arginine, l-Citruline, Fetal growth, percentile,
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: Clinical Trial open controlled parallel randomized simple
Who Masked: Participant, Investigator
Masking Description: we don´t know who receives the intervention and who receives the placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental L-arginine 3 g and L-citruline 2 g (Experimental): Drug: L-arginine 3g and L-citruline 2g, Food supplement, PO , for 24 h, until birth
  Interventions: Dietary Supplement: L-arginine 3g + L-Citruline 2 g
- placebo (Experimental): Placebo 3g ( starch ) PO for 24 h. until birth
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine 3g + L-Citruline 2 g — receive L-arginine 3g + l-Citruline 2 g PO, for 24 h, until birth.
  Other Names: L-arginine 3g; L-Citruline 2 g
  Arms: Experimental L-arginine 3 g and L-citruline 2 g
Drug: Placebo — receive placebo 3g PO, for 24 h, until birth.
  Arms: placebo

SUMMARY:
Introduction:

The high incidence of intrauterine growth restriction is a public health problem; in this pathology, newborns present weight below the 10th percentile, this implies an increase in morbidity in the short term (complications due to hypoxia) and long term (pathologies typical of Fetal Programming) as well as the cost of health services. L-arginine at different doses has been used for some pathologies such as preeclampsia with controversial results. Authors have mentioned that the joint administration of l-citrulline can increase the efficacy of l-arginine. A stunted fetus is a challenge for the fetal physician; due to the complexity of the follow-up, but above all to determine the moment for the termination of the pregnancy. Finding some treatment to promote weight gain would improve the short- and long-term expectations of these infants.

General objective To determine the efficacy of L-arginine + L-Citrulline (3 / 2g) every 24 hours, in fetuses with a decrease in their growth curve in the third trimester of pregnancy.

Material and methods Clinical trial, parallel, controlled, randomized simple, Double blind. Two groups of pregnant women will be carried out in the third trimester; fetus with a decrease in its growth curve, percentile> 10 and <25 for gestation age, they will be given an informed consent letter and they will be randomized (double blind), they will proceed to give intervention (L-arginine + Citrin (3 / 2 g) every 24 hours Vs placebo), a follow-up will be carried out every two weeks, where the weight and growth curve will be calculated in percentile, until the resolution of the pregnancy and data will be taken from the perinatal results in both groups.

Statistic analysis Medics of central tendency will be calculated and Chi squared will be applied for qualitative variables, T of student for qualitative variables and it is considered P <0.005.

DETAILED DESCRIPTION:
50 patients with a pregnancy of more than 26 weeks of gestation, 25 with intervention and 25 control will be included; in which the fetus is between 10 and 25th percentile . It will be carried out in the obstetric service of the old civil hospital, with a double-blind randomization.

Evaluations will be carried out every two weeks where the fetal weight, umbilical artery Doppler, middle cerebral artery, venous duct, uterine arteries, amniotic fluid, placenta will be evaluated.

The assessment will be made until birth, from where the birth weight, height, Apgar, Capurro score, characteristics and placental weight, approximate bleeding will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy with a single fetus
* Patient over 18 years of age
* Patient under 35 years of age
* Pregnancy greater than 25 weeks' gestation confirmed by first trimester ultrasound or reliable last period
* Fetus with decrease or flattening of its growth curve by ultrasound (P> 10 and <25)
* Apparently healthy fetus
* Fetus without Doppler alterations in any of its blood vessels (Venous Ductus, Cerebral Artery medial, Umbilical Artery .

Exclusion Criteria:

* Fetus diagnosed with a malformation
* Fetus diagnosed with a syndrome or chromosomopathy
* Fetus below the 10th percentile for gestational age by ultrasound
* Mother with Type 1, Type 2 or Gestational Diabetes mellitus.
* Chronic maternal hypertension
* Preeclampsia with data of severity or early onset
* Aspirin intake (100-150 mg a day from the first trimester of pregnancy)
* Fetus with a poor ultrasonographic window for evaluation.
* Mother with BMI <18.5 prior to pregnancy
* Maternal BMI> 30
* Known allergy to treatment
* Non-reassuring fetal state.
* Abnormal placental insertion.
* Patient with renal insufficiency, LUPUS or Antiphospholipid syndrome

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — single pregnancy in third trimester with fetus between the 10th to 25th percentile
Enrollment: 41 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2021-10-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Fetal Growth | 10 weeks
  fetal weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Milton Omar Guzman Ornelas, Dr., Study Director — University of Guadalajara

REFERENCES:
- [Background] Dover GJ. The Barker hypothesis: how pediatricans will diagnose and prevent common adult-onset diseases. Trans Am Clin Climatol Assoc. 2009;120:199-207. No abstract available. PMID 19768178
- [Result] Ananth CV, Vintzileos AM. Distinguishing pathological from constitutional small for gestational age births in population-based studies. Early Hum Dev. 2009 Oct;85(10):653-8. doi: 10.1016/j.earlhumdev.2009.09.004. Epub 2009 Sep 27. PMID 19786331
- [Result] Barker DJ, Osmond C, Kajantie E, Eriksson JG. Growth and chronic disease: findings in the Helsinki Birth Cohort. Ann Hum Biol. 2009 Sep-Oct;36(5):445-58. doi: 10.1080/03014460902980295. PMID 19562567
- [Result] Bourdon A, Parnet P, Nowak C, Tran NT, Winer N, Darmaun D. L-Citrulline Supplementation Enhances Fetal Growth and Protein Synthesis in Rats with Intrauterine Growth Restriction. J Nutr. 2016 Mar;146(3):532-41. doi: 10.3945/jn.115.221267. Epub 2016 Feb 10. PMID 26865647
- [Result] Bujold E, Morency AM, Roberge S, Lacasse Y, Forest JC, Giguere Y. Acetylsalicylic acid for the prevention of preeclampsia and intra-uterine growth restriction in women with abnormal uterine artery Doppler: a systematic review and meta-analysis. J Obstet Gynaecol Can. 2009 Sep;31(9):818-826. doi: 10.1016/S1701-2163(16)34300-6. PMID 19941706
- [Result] Byrne BM, Howard RB, Morrow RJ, Whiteley KJ, Adamson SL. Role of the L-arginine nitric oxide pathway in hypoxic fetoplacental vasoconstriction. Placenta. 1997 Nov;18(8):627-34. doi: 10.1016/s0143-4004(97)90003-5. PMID 9364597
- [Result] Camarena Pulido EE, Garcia Benavides L, Panduro Baron JG, Pascoe Gonzalez S, Madrigal Saray AJ, Garcia Padilla FE, Totsuka Sutto SE. Efficacy of L-arginine for preventing preeclampsia in high-risk pregnancies: A double-blind, randomized, clinical trial. Hypertens Pregnancy. 2016 May;35(2):217-25. doi: 10.3109/10641955.2015.1137586. Epub 2016 Mar 22. PMID 27003763
- [Result] Chen J, Gong X, Chen P, Luo K, Zhang X. Effect of L-arginine and sildenafil citrate on intrauterine growth restriction fetuses: a meta-analysis. BMC Pregnancy Childbirth. 2016 Aug 16;16:225. doi: 10.1186/s12884-016-1009-6. PMID 27528012
- [Result] Colella M, Frerot A, Novais ARB, Baud O. Neonatal and Long-Term Consequences of Fetal Growth Restriction. Curr Pediatr Rev. 2018;14(4):212-218. doi: 10.2174/1573396314666180712114531. PMID 29998808
- [Result] Cottrell E, Tropea T, Ormesher L, Greenwood S, Wareing M, Johnstone E, Myers J, Sibley C. Dietary interventions for fetal growth restriction - therapeutic potential of dietary nitrate supplementation in pregnancy. J Physiol. 2017 Aug 1;595(15):5095-5102. doi: 10.1113/JP273331. Epub 2017 Feb 27. PMID 28090634
- [Result] Crispi F, Miranda J, Gratacos E. Long-term cardiovascular consequences of fetal growth restriction: biology, clinical implications, and opportunities for prevention of adult disease. Am J Obstet Gynecol. 2018 Feb;218(2S):S869-S879. doi: 10.1016/j.ajog.2017.12.012. PMID 29422215